CLINICAL TRIAL: NCT03113968
Title: ELEKT-D: Electroconvulsive Therapy (ECT) vs. Ketamine in Patients With Treatment Resistant Depression (TRD)
Acronym: ELEKT-D
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bo Hu (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Bo Hu, Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELEKT-D
Record Dates: First submitted 2017-02-09; First posted 2017-04-14 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Treatment Resistant Depression; Electroconvulsive Therapy; ECT; Ketamine; Psychiatric Disorder; Depression; Major Depressive Disorder; Major Depressive Episode; Unipolar Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Mental Disorders; Depression; Depressive Disorder, Major; Depressive Disorder | interventions — Electroconvulsive Therapy; Ketamine

STUDY DESIGN:
Intervention Model Description: unblinded prospective randomized open-label
Masking Description: Due to the nature of the study treatments it is not possible to blind patients or investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- electroconvulsive therapy (ECT) (Active Comparator): Treatments will be given 3 times a week up to a total of 9 treatments over 3 - 5 weeks. Initial ECT treatment is Right Unilateral (RUL) ultra-brief pulse at 6X seizure threshold. Seizure threshold and dose can be increased per investigator and patient discretion.
  Interventions: Procedure: electroconvulsive therapy (ECT)
- ketamine infusion (Active Comparator): Treatments will be given 2 times a week up to a total of 6 treatment over 3 - 5 weeks. Initial standard dose will be 0.5 mg/kg infusion over 40 min. The dose can be modified if clinically warranted per investigator and patient discretion.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Procedure: electroconvulsive therapy (ECT) — ECT is a procedure done under general anesthesia where small electric currents are passed through the brain, intentionally triggering a brief seizure. Patients who have not responded to antidepressant medications may be candidates for ECT. ECT is FDA approved for treatment resistant depression.
  Arms: electroconvulsive therapy (ECT)
Drug: Ketamine — Ketamine is a medication that is used as a short acting anesthetic in pediatric and adult medicine. Subanesthetic (low) doses will be given to patients via infusion in order to assess whether it helps with depression symptoms in patients who have not responded to antidepressant therapy. Ketamine is not FDA approved for this indication and its effectiveness in treatment resistant depression has not been proven. Prior studies have indicated that subanesthetic doses of ketamine may be helpful for treatment resistant depression.
  Arms: ketamine infusion

SUMMARY:
The goal of the study is to conduct a comparative randomized trial of electroconvulsive therapy (ECT) vs. ketamine for patients with treatment resistant depression (TRD) in a real world setting with patient reported outcomes as primary and secondary outcome measures.

DETAILED DESCRIPTION:
Patients with treatment resistant depression who meet all inclusion criteria and do not meet any exclusion criteria will be randomized to either electroconvulsive therapy (ECT) three times per week or ketamine infusion two times per week. Patients will answer questionnaires about their symptoms prior to treatments. The acute treatment phase of the study will last three to five weeks. Depending on response to treatment, some patients will be followed for an additional six months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any study related procedures are performed
2. Inpatients or outpatients referred by their providers for ECT treatment and eligible for ECT treatment
3. Males/females at least 21 years of age but no older than 75 years of age
4. Meet DSM-5 criteria for Major Depressive Episode as determined by both:

   A. a clinician's diagnostic evaluation and B. confirmed with the MINI International Neuropsychiatric Interview (MINI 7.0.2)
5. A current depressive episode that has lasted a minimum of 4 weeks
6. Meet all of the following criteria on symptom rating scales at screening:

   A. Montgomery Asberg Depression Rating Scale (MADRS) score >20 B. Young Mania Rating Scale (YMRS) of ≤ 5 C. Montreal Cognitive Assessment (MoCA) of ≥18
7. Have had ≥2 adequate trials of antidepressants or augmentation strategies during their lifetime. An adequate trial is defined as 4 weeks of medication at the minimum FDA approved dose. This will be equal to a trial rating of 3 or more.
8. In the opinion of the investigator, the patient is willing and able to comply with scheduled visits, treatment plan, and other trial procedures for the duration of the study

Exclusion Criteria:

1. Meet DSM-5 criteria for bipolar disorder, schizophrenia, schizophreniform disorder, schizoaffective disorder, mental retardation, or pervasive developmental disorder
2. Meets any exclusion criteria for ECT or ketamine treatment as described in the clinical guidelines or according to investigator judgment
3. The patient is pregnant or breast feeding
4. The patient has a severe medical illness or severe neurological disorder
5. The patient has a known ketamine allergy or is taking a medication that may interact with ketamine
6. Diagnosis of major depressive disorder with psychotic features during the current depressive episode
7. Unable to give informed consent
8. Was previously enrolled/randomized into the trial

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — The Cleveland Clinic
Locations (5):
- United States (5):
  - Yale School of Medicine, New Haven, Connecticut
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nemeroff CB. Prevalence and management of treatment-resistant depression. J Clin Psychiatry. 2007;68 Suppl 8:17-25. PMID 17640154
- [Background] Kellner CH, Greenberg RM, Murrough JW, Bryson EO, Briggs MC, Pasculli RM. ECT in treatment-resistant depression. Am J Psychiatry. 2012 Dec;169(12):1238-44. doi: 10.1176/appi.ajp.2012.12050648. PMID 23212054
- [Background] Lisanby SH. Electroconvulsive therapy for depression. N Engl J Med. 2007 Nov 8;357(19):1939-45. doi: 10.1056/NEJMct075234. No abstract available. PMID 17989386
- [Background] Newport DJ, Carpenter LL, McDonald WM, Potash JB, Tohen M, Nemeroff CB; APA Council of Research Task Force on Novel Biomarkers and Treatments. Ketamine and Other NMDA Antagonists: Early Clinical Trials and Possible Mechanisms in Depression. Am J Psychiatry. 2015 Oct;172(10):950-66. doi: 10.1176/appi.ajp.2015.15040465. PMID 26423481
- [Background] Sanacora G, Heimer H, Hartman D, Mathew SJ, Frye M, Nemeroff C, Robinson Beale R. Balancing the Promise and Risks of Ketamine Treatment for Mood Disorders. Neuropsychopharmacology. 2017 May;42(6):1179-1181. doi: 10.1038/npp.2016.193. Epub 2016 Sep 19. No abstract available. PMID 27640324
- [Derived] Kumpf KT, Wilkinson ST, Hu B, Chen R, Krishnan K, Chakrabarti S, Rhee TG, Grezmak T, Mathew SJ, Sanacora G, Murrough JW, Goes FS, Collins KA, Barnett BS, Anand A. Comparing the Cognitive Effects of Repeated Intravenous Ketamine and Electroconvulsive Therapy in Patients With Treatment-Resistant Depression: A Secondary Analysis of the ELEKT-D Trial. J Clin Psychiatry. 2025 Sep 3;86(4):25m15781. doi: 10.4088/JCP.25m15781. PMID 40900112
- [Derived] Anand A, Mathew SJ, Sanacora G, Murrough JW, Goes FS, Altinay M, Aloysi AS, Asghar-Ali AA, Barnett BS, Chang LC, Collins KA, Costi S, Iqbal S, Jha MK, Krishnan K, Malone DA, Nikayin S, Nissen SE, Ostroff RB, Reti IM, Wilkinson ST, Wolski K, Hu B. Ketamine versus ECT for Nonpsychotic Treatment-Resistant Major Depression. N Engl J Med. 2023 Jun 22;388(25):2315-2325. doi: 10.1056/NEJMoa2302399. Epub 2023 May 24. PMID 37224232
- [Derived] Mathew SJ, Wilkinson ST, Altinay M, Asghar-Ali A, Chang LC, Collins KA, Dale RM, Hu B, Krishnan K, Kellner CH, Malone DA, Murrough JW, Ostroff RB, Sanacora G, Shao M, Anand A. ELEctroconvulsive therapy (ECT) vs. Ketamine in patients with Treatment-resistant Depression: The ELEKT-D study protocol. Contemp Clin Trials. 2019 Feb;77:19-26. doi: 10.1016/j.cct.2018.12.009. Epub 2018 Dec 17. PMID 30572160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2017 - September 2022, outpatients or inpatients referred by their clinical providers to a site's ECT service for treatment were invited to participate in the study. Patients suffering from TRD who were interested in participation were enrolled after providing written informed consent.
Pre-assignment Details: Of 2321 patients assessed, 436 met the inclusion criteria and were screened. 33 had screen failures and 403 were randomized.
Period: Overall Study
Arm/Group | Electroconvulsive Therapy (ECT) | Ketamine Infusion
Started | 203 | 200
Completed | 172 | 196
Not Completed | 31 | 4
Not completed — Withdrawal by Subject | 31 | 4

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Electroconvulsive Therapy (ECT) | Ketamine Infusion | Total
Number analyzed (Participants) | 203 | 200 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.1) | 45.6 (14.8) | 46.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 106 | 206
  Male | 103 | 94 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 24 | 35
  Not Hispanic or Latino | 192 | 176 | 368
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 182 | 173 | 355
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (7.9) | 29.5 (7.4) | 29.9 (7.6)
Inpatient at first treatment [Count of Participants; unit: Participants] | 21 | 23 | 44
Age of onset of First Major Depression - yrs [Mean (Standard Deviation); unit: years] | 19.4 (11) | 19.7 (11.5) | 19.5 (11.2)
Number of Past Major Depression Episodes [Median (Inter-Quartile Range); unit: Episodes] | 5 [2 to 18] | 5 [2 to 16] | 5 [2 to 16]
Duration of Current Episode - month [Median (Inter-Quartile Range); unit: months] | 24 [10 to 72] | 24 [10 to 75] | 24 [10 to 72]
Number of Patients with Family History of Depression [Count of Participants; unit: Participants] | 160 | 154 | 314
Attempted Suicide [Count of Participants; unit: Participants] | 84 | 73 | 157
Previous ECT [Count of Participants; unit: Participants] | 21 | 23 | 44
Previous Ketamine [Count of Participants; unit: Participants] | 8 | 14 | 22
16-item Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) [Mean (Standard Deviation); unit: units on a scale] — Score ranges from 0 to 27 with higher scores indicating greater depression
  units on a scale | 18.2 (4.2) | 17.9 (4.1) | 18.1 (4.1)
Montgomery-Åsberg Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 0 to 60 with higher scores indicating greater depression
  units on a scale | 32.6 (6) | 32.3 (6.2) | 32.5 (6.1)
Clinical Global Impression-Severity (CGI-S) scale [Mean (Standard Deviation); unit: units on a scale] — Scale ranges from 1 to 7, with higher scores indicating more severe depression
  units on a scale | 5.2 (0.6) | 5.0 (0.6) | 5.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Responses Based on the 16-item Quick Inventory of Depressive Symptomatology-Self-Report Scale (QIDS-SR-16)
Description: Response is defined as at least a 50% improvement in the QIDS-SR-16 scale from baseline to the End of Treatment visit. The End of Treatment visit will occur 3-5 weeks after the Baseline visit.
Time Frame: Acute Study Phase (Baseline Visit to End of Treatment Visit) - approximately 3-5 weeks
Population: Modified Intention-to-treat Population (i.e., participants with at least one treatment and at least one follow-up measurement)
Measure: Count of Participants; unit: Participants
Arm/Group | Electroconvulsive Therapy (ECT) | Ketamine Infusion
Number analyzed (Participants) | 170 | 195
Participants | 70 | 108
Statistical Analysis 1: Comparison: Electroconvulsive Therapy (ECT) vs Ketamine Infusion; Test type: Non-Inferiority — The Farrington-Manning score test was used to assess the noninferiority of KET; p < .001, The Farrington-Manning score test

2. Secondary Outcome: Number of Participants With Treatment Responses Based on the Montgomery-Åsberg Rating Scale (MADRS)
Description: The outcome measure was the percentage of responders at the end-of-treatment visit, defined as a ≥50% decrease in MADRS score from the baseline visit (i.e., first treatment visit) to the end-of-treatment visit (within 3 days of last treatment).
Time Frame: Acute Study Phase (Baseline Visit to End of Treatment Visit) - approximately 3-5 weeks
Population: Modified intention-to-treat population (i.e., participants with at least one treatment and at least one follow-up measurement). One participant in the ECT group had missing baseline MADRS and was further excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Electroconvulsive Therapy (ECT) | Ketamine Infusion
Number analyzed (Participants) | 169 | 195
Participants | 70 | 99
Statistical Analysis 1: Comparison: Electroconvulsive Therapy (ECT) vs Ketamine Infusion; Test type: Superiority; Mean Difference (Net) = 9.3; P-values not reported

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the period from baseline to the end-of-treatment visit (up to 5 weeks from baseline)
Description: Adverse events were reported for the modified Intention-to-Treat population (participants who received at least one treatment and had at least follow-up measurement). The subset of treatment responders in both groups were followed for an observational period of additional six months, and during this period these participants might be on different treatments as clinically needed.
Arm/Group | Electroconvulsive Therapy (ECT) | Ketamine Infusion
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/195
Serious Adverse Events (participants affected / at risk) | 4/170 | 5/195
Other Adverse Events (participants affected / at risk) | 27/170 | 32/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electroconvulsive Therapy (ECT) (N=170) | Ketamine Infusion (N=195)
Chest pain (Cardiac disorders) | 0 | 1
Infection requiring antibiotics (Infections and infestations) | 1 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0
Aborted suicide attempt (gesture) (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 3
Asystole (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Electroconvulsive Therapy (ECT) (N=170) | Ketamine Infusion (N=195)
Headache (General disorders) | 12 | 16
Hypertension (severe / prolonged) (Cardiac disorders) | 4 | 6
Muscle Pain / Weakness (Musculoskeletal and connective tissue disorders) | 9 | 1
Nausea (Gastrointestinal disorders) | 6 | 10
Non-Cardiac Jaw Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Panic (Psychiatric disorders) | 3 | 4
Suicidal Ideation (Psychiatric disorders) | 2 | 4

LIMITATIONS AND CAVEATS:
Our trial has several limitations. ECT was started with right unilateral placement and was then switched to bilateral placement in the event of inadequate response. The open-label design of our trial could have influenced response. Maintenance treatment was not studied. Other limitations of our trial include a lack of placebo, the flexibility of treatment methods, and a follow-up period during which the patients received treatment as presc

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03113968/Prot_001.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03113968/SAP_002.pdf